CLINICAL TRIAL: NCT01054469
Title: Ultrasound Guided Transversus Abdominus Plane Block for Patients Undergoing Laparoscopic Hand-assisted Nephrectomy.
Brief Title: Transversus Abdominus Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Stephen Aniskevich, III, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 08-003563
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Nephrectomy
Keywords: nephrectomy
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block with placebo (Placebo Comparator)
  Interventions: Procedure: TAP block placement with placebo
- TAP block with ropivacaine (Active Comparator)
  Interventions: Procedure: Placement of block with ropivacaine

INTERVENTIONS:
Procedure: TAP block placement with placebo — 20 ml of normal saline (placebo)
  Arms: TAP block with placebo
Procedure: Placement of block with ropivacaine — 20 ml of 0.5% ropivacaine hydrochloride
  Arms: TAP block with ropivacaine

SUMMARY:
Transversus Abdominus Plane (TAP) block may reduce need for postoperative pain medications in patients undergoing laparoscopic hand assisted nephrectomy. Our hypothesis is that the TAP block will result in a significant reduction in pain scores and morphine requirements in the active group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥ 18 and ≤ 80 years of age.
* Patients scheduled to undergo hand assisted laparoscopic removal of a single kidney for either tumor or living donor transplantation.

Exclusion Criteria:

* Patients scheduled to undergo an open procedure for nephrectomy
* Patients who are converted from hand assisted laparoscopic surgery to open surgery due to intraoperative complications.
* Bilateral nephrectomy
* Pregnant or lactating patients
* Patients unable or unwilling to provide informed consent
* Patients unable to comprehend the use of a visual analog scale
* Patients desiring preemptive antiemetics
* Opioid tolerance
* Allergy to amide local anesthetics or any of the study drugs (morphine).
* Contraindication to regional nerve block (bleeding disorder, infection at site of block)
* Patients with history of dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Determine if TAP block is a viable alternative to PCA narcotics for the control of pain after hand-assisted, laparoscopic nephrectomy. | 24 hours postoperatively

SECONDARY OUTCOMES:
TAP block with ropivacaine will lead to equivalent or better results with regard to the following outcomes:pain scores, nausea, vomiting, sedation, request for PCA, discontinuation of Foley catheter, discharge from the hospital | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Aniskevich, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States